CLINICAL TRIAL: NCT00220415
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel Group Trial to Investigate the Efficacy and Safety of SPM 927 (200mg/Day and 400mg/Day) as Adjunctive Therapy in Subjects With Partial Seizures With or Without Secondary Generalization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0755; 2004-000290-58 (EudraCT Number)
Record Dates: First submitted 2005-08-30; First posted 2005-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2010-02

CONDITIONS: Partial Seizures With or Without Secondary Generalization
MeSH Terms: interventions — 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

INTERVENTIONS:
Drug: SPM 927

SUMMARY:
Male and female patients between 16 and 70 years of age who are diagnosed with epilepsy with partial seizures and are taking up to 3 medications for this medical condition will take part in this research study at approximately 80 different locations in Australia and Europe.

The purpose of this study is to evaluate the effectiveness, safety and tolerability of consistent dosages of study drug (lacosamide) taken orally twice a day for about 4 months.

Each patient who qualifies and chooses to participate in the study will receive placebo (inactive drug) or gradually increasing doses of lacosamide (SPM 927) up to the target dose of 200mg/day or 400mg/day. The target dose or placebo will be maintained for 12 weeks.

The study clinic visits will include a medical history and physical exam, ECG, blood and urine sample collection, and completion of a seizure diary.

Patients who complete the study may enroll in an extension trial and receive active study drug.

ELIGIBILITY:
Inclusion Criteria:

* partial seizures with or without secondary generalization

Exclusion Criteria:

* subjects received SPM 927 in a previous trial

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-05; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, Monheim, Germany

REFERENCES:
- [Result] Halasz P, Kalviainen R, Mazurkiewicz-Beldzinska M, Rosenow F, Doty P, Hebert D, Sullivan T; SP755 Study Group. Adjunctive lacosamide for partial-onset seizures: Efficacy and safety results from a randomized controlled trial. Epilepsia. 2009 Mar;50(3):443-53. doi: 10.1111/j.1528-1167.2008.01951.x. Epub 2009 Jan 17. PMID 19183227
- [Result] Sake JK, Hebert D, Isojarvi J, Doty P, De Backer M, Davies K, Eggert-Formella A, Zackheim J. A pooled analysis of lacosamide clinical trial data grouped by mechanism of action of concomitant antiepileptic drugs. CNS Drugs. 2010 Dec;24(12):1055-68. doi: 10.2165/11587550-000000000-00000. PMID 21090839
- [Result] Borghs S, de la Loge C, Cramer JA. Defining minimally important change in QOLIE-31 scores: estimates from three placebo-controlled lacosamide trials in patients with partial-onset seizures. Epilepsy Behav. 2012 Mar;23(3):230-4. doi: 10.1016/j.yebeh.2011.12.023. Epub 2012 Feb 15. PMID 22341962
- [Derived] Biton V, Gil-Nagel A, Isojarvi J, Doty P, Hebert D, Fountain NB. Safety and tolerability of lacosamide as adjunctive therapy for adults with partial-onset seizures: Analysis of data pooled from three randomized, double-blind, placebo-controlled clinical trials. Epilepsy Behav. 2015 Nov;52(Pt A):119-27. doi: 10.1016/j.yebeh.2015.09.006. Epub 2015 Sep 27. PMID 26414341